CLINICAL TRIAL: NCT03439345
Title: A Randomised Placebo-controlled Trial of Fenofibrate to Prevent Progression of Non-proliferative Retinopathy in Diabetes
Brief Title: Lowering Events in Non-proliferative Retinopathy in Scotland
Acronym: LENS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Glasgow (Other); University of Aberdeen (Other); University of Dundee (Other); University of Edinburgh (Other); NHS Scotland Diabetic Retinopathy Screening Collaborative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTSULENS1; ISRCTN15073006 (Registry Identifier: International Standard Randomised Controlled Trial Number)
Record Dates: First submitted 2018-02-05; First posted 2018-02-20 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fenofibrate 145 mg (Experimental): Name: Fenofibrate; Form: tablet; Dosage: 145 mg; Frequency: One tablet (taken daily with normal renal function, taken every second day with chronic kidney disease)
  Interventions: Drug: Fenofibrate 145 mg
- Placebo Oral Tablet (Placebo Comparator): Name: Placebo; Form: tablet; Dosage: not applicable; Frequency: One tablet (taken daily with normal renal function, taken every second day with chronic kidney disease)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Fenofibrate 145 mg — One tablet (taken daily with normal renal function, taken every second day with chronic kidney disease)
  Arms: Fenofibrate 145 mg
Drug: Placebo Oral Tablet — One tablet (taken daily with normal renal function, taken every second day with chronic kidney disease)
  Arms: Placebo Oral Tablet

SUMMARY:
LENS is a streamlined multicentre randomised placebo-controlled parallel-group trial investigating the effect of fenofibrate treatment on the progression of diabetic retinopathy/maculopathy.

DETAILED DESCRIPTION:
LENS is a phase 4 randomised placebo-controlled clinical trial of fenofibrate in participants with diabetes and observable retinopathy or maculopathy. The trial aims to recruit approximately 1,060 participants and to treat them for a median duration of at least 4 years. The main aim of LENS is to investigate the effect of fenofibrate therapy on progression to referable diabetic retinopathy/maculopathy. The trial will be conducted using a pragmatic streamlined trial design with the only planned face-to-face visits being an initial screening visit, followed by a randomisation visit eight weeks later. Contact with participants thereafter will be by means of regular telephone or computer questionnaire, and outcome and safety data will also be sought by means of linkage to NHS Scotland registries. Prior to randomisation, eligible participants will enter an active run-in phase of 6 to 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving informed consent
2. Diabetes Mellitus (any type except gestational diabetes)
3. Observable diabetic retinopathy/maculopathy (defined based on NHS Scotland grading criteria as: R1 in both eyes or R2 in one/both eyes at the most recent retinal screening assessment; or M1 in one/both eyes at any retinal screening assessment in the 3 years)
4. Willing to either complete electronic questionnaires or conduct telephone interviews for collection of data once every 6 months

Exclusion Criteria:

1. Clinically significant DR (defined as R3 or R4 or M2 in one or both eyes)
2. History of gallbladder disease (cholecystitis, symptomatic gallstones, cholecystectomy)
3. History of acute or chronic pancreatitis
4. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2X the upper limit of normal (ULN) according to local NHS laboratory reference range at screening visit
5. ALT or AST >2.5X ULN according to local NHS laboratory reference range at randomisation visit
6. Creatine kinase (CK) >3X ULN according to local NHS laboratory reference range at screening visit
7. CK >3X ULN according to local NHS laboratory reference range at randomisation visit
8. Estimated glomerular filtration rate (eGFR) <40mL/min/1.73m2 at screening visit
9. eGFR <30mL/min/1.73m2 at randomisation visit
10. Cirrhosis of any aetiology or any other serious hepatic disease (investigator opinion)
11. Female who is pregnant, breastfeeding, currently trying to become pregnant, or of child-bearing potential and not practising birth control
12. Ongoing vitamin K antagonist (warfarin, phenindione, acenocoumarol), cyclosporine, colchicine, ketoprofen, daptomycin, fibrate therapy, or treatment with rosuvastatin 40mg daily
13. Previous myositis, myopathy or rhabdomyolysis of any cause, or diagnosed hereditary muscle disorder
14. Ongoing renal replacement therapy
15. Any previous organ transplant
16. Previous reported intolerance to any fibrate
17. Medical history that might limit the individual's ability to take trial treatments for the duration of the study (e.g. severe respiratory disease, history of cancer within last 5 years other than non-melanoma skin cancer; or recent history of alcohol or substance misuse)
18. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial
19. LENS participants can participate in other research studies, including clinical trials. The only exclusions related to co-enrolment will be: if any other study or trial excludes co-enrolment or if the intervention being investigated in another trial has the potential to interact with fenofibrate therapy.
20. Not adherent to active run-in treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1151 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Preiss, PhD FRCPath, Principal Investigator — University of Oxford
Locations (16):
- United Kingdom (16):
  - NHS Grampian, Aberdeen
  - NHS Lanarkshire, Airdrie
  - NHS Ayrshire and Arran, Ayr
  - NHS Dumfries and Galloway, Dumfries
  - NHS Tayside, Dundee
  - NHS Fife, Dunfermline
  - NHS Lanarkshire, East Kilbride
  - NHS Lothian, Edinburgh
  - NHS Greater Glasgow and Clyde, Glasgow
  - NHS Highland, Inverness
  - NHS Ayrshire and Arran, Kilmarnock
  - NHS Fife, Kirkcaldy
  - NHS Forth Valley, Larbert
  - NHS Borders, Melrose
  - NHS Tayside, Perth
  - NHS Lanarkshire, Wishaw

IPD SHARING:
Plan to Share IPD: Yes
Data generated by LENS will be available on application to bona fide academic researchers in accordance with the Data Access Policy for the Nuffield Department of Population Health, University of Oxford. Such approvals will also need to be consistent with the informed consent provided by participants. Any sharing of data derived from NHS Scotland data will need to comply with the approvals of the trial.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Applications will be considered in accordance with Data Access Policy for the Nuffield Department of Population Health, University of Oxford.
URL: https://www.ndph.ox.ac.uk/files/about/ndph-data-access-policy-1.pdf

REFERENCES:
- [Background] LENS Collaborative Group. Design, recruitment and baseline characteristics of the LENS trial. Diabet Med. 2024 Sep;41(9):e15310. doi: 10.1111/dme.15310. Epub 2024 Feb 22. PMID 38385587
- [Result] Preiss D, Logue J, Sammons E, Zayed M, Emberson J, Wade R, Wallendszus K, Stevens W, Cretney R, Harding S, Leese G, Currie G, Armitage J. Effect of Fenofibrate on Progression of Diabetic Retinopathy. NEJM Evid. 2024 Aug;3(8):EVIDoa2400179. doi: 10.1056/EVIDoa2400179. Epub 2024 Jun 21. PMID 38905569
- See also: LENS trial website — https://www.ctsu.ox.ac.uk/lens

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Started | 576 | 575
Completed | 576 | 573
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Consent withdrawn | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet | Total
Number analyzed (Participants) | 576 | 575 | 1151
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age at randomisation
  years | 60.8 (12.4) | 60.6 (12.3) | 60.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156 | 156 | 312
  Male | 420 | 419 | 839
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 567 | 558 | 1125
  Other | 4 | 9 | 13
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — All patients enrolled were from Scotland
  participants
    United Kingdom | 576 | 575 | 1151
Type of diabetes mellitus [Count of Participants; unit: Participants]
  Type 1 | 154 | 151 | 305
  Type 2 | 421 | 423 | 844
  Other | 1 | 1 | 2
Duration of diabetes [Mean (Standard Deviation); unit: years] | 18.3 (10.5) | 17.7 (10.0) | 18 (10.25)
Retinopathy grading (worse grade) [Count of Participants; unit: Participants] — Worse eye retinopathy defined as R2>R1>R0. Retinopathy was graded according to NHS Scotland's Diabetic Eye Screening Programme grading scheme. R1 (mild background diabetic retinopathy): the presence of at least one of any of the following features: dot hemorrhages / microaneurysms, hard exudates, cotton wool spots, blot hemorrhages, superficial/ flame shaped hemorrhages). R2 (observable background retinopathy): four or more blot haemorrhages in one hemi-field only (inferior and superior hemi-fields delineated by a line passing through the centre of the fovea and optic disc).
  Participants
    No retinopathy (R0) | 5 | 4 | 9
    Mild background retinopathy (R1) | 562 | 564 | 1126
    Observable background retinopathy (R2) | 9 | 7 | 16
Maculopathy grading (worse eye) [Count of Participants; unit: Participants] — Worse eye maculopathy was defined as M1 > M0. Maculopathy was graded according to NHS Scotland's Diabetic Eye Screening Programme grading scheme. M1 (observable maculopathy): hard exudates within a radius of >1 but ≤2 optic disc diameters from the centre of the fovea.
  Participants
    No maculopathy (M0) | 517 | 515 | 1032
    Observable diabetic maculopathy (M1) | 59 | 60 | 119
Retinal laser treatment or intravitreal injections or vitrectomy [Count of Participants; unit: Participants] | 53 | 59 | 112
Cardiovascular disease [Count of Participants; unit: Participants] | 103 | 96 | 199
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] — Based on measurements at the randomisation assessment. Population: Blood pressure data missing for 70 participants
  mm Hg
    number analyzed (Participants) | 542 | 539 | 1081
    (all) | 136.7 (17.2) | 136.4 (17.9) | 136.6 (17.5)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] — Based on measurements at the randomisation assessment. Population: Blood pressure data missing for 70 participants
  mm Hg
    number analyzed (Participants) | 542 | 539 | 1081
    (all) | 75.4 (9.4) | 75.5 (9.3) | 75.5 (9.4)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Based on measurements at the randomisation assessment. The body-mass index is the weight in kilograms divided by the square of the height in meters. Population: Body mass index data missing for 35 participants.
  kg/m^2
    number analyzed (Participants) | 559 | 557 | 1116
    (all) | 30.9 (6.4) | 30.7 (6.0) | 30.8 (6.2)
Haemoglobin A1C (HbA1c): [Mean (Standard Deviation); unit: mmol/mol] — Based on blood tests at the screening assessment. Population: HbA1c data missing for 74 participants.
  mmol/mol
    number analyzed (Participants) | 538 | 539 | 1077
    (all) | 66.4 (16.1) | 66.3 (15.9) | 66.4 (16.0)
Creatinine at Screening [Mean (Standard Deviation); unit: mg/dl] | 0.88 (0.21) | 0.88 (0.21) | 0.88 (0.21)
Creatinine at Randomisation [Mean (Standard Deviation); unit: mg/dl] | 1.01 (0.26) | 1.00 (0.25) | 1.01 (0.25)
Estimated Glomerular Filtration Rate (eGFR) at Screening [Count of Participants; unit: Participants]
  <60ml/min/1.73 m^2 | 58 | 40 | 98
  ≥60ml/min/1.73 m^2 | 518 | 535 | 1053
Estimated Glomerular Filtration Rate (eGFR) at Randomisation [Count of Participants; unit: Participants]
  <60 ml/min/1.73 m^2 | 130 | 131 | 261
  ≥60 ml/min/1.73 m^2 | 446 | 444 | 890
Total cholesterol (mg/dl) [Mean (Standard Deviation); unit: mg/dl] — Based on blood tests at the screening assessment. Population: Total cholesterol data missing for 12 participants.
  mg/dl
    number analyzed (Participants) | 572 | 567 | 1139
    (all) | 156 (37) | 157 (38) | 156.5 (37.5)
HDL cholesterol (mg/dl) [Mean (Standard Deviation); unit: mg/dl] — Based on blood tests at the screening assessment. Population: HDL cholesterol data missing for 23 participants.
  mg/dl
    number analyzed (Participants) | 568 | 560 | 1128
    (all) | 51 (16) | 50 (15) | 50.5 (15.5)
Triglycerides (IQR) (mg/dl) [Median (Inter-Quartile Range); unit: mg/dl] — Based on blood tests at the screening assessment. Triglycerides are shown as median (interquartile range [IQR]) Population: Triglyceride data missing for 17 participants.
  mg/dl
    number analyzed (Participants) | 571 | 563 | 1134
    (all) | 137 [90 to 205] | 138 [97 to 195] | 137 [94 to 202]
Baseline medications [Number; unit: participants]
  Non-insulin glucose-lowering therapy | 396 | 389 | 785
  Insulin | 256 | 249 | 505
  Statin | 425 | 429 | 854
  Renin-angiotensin system inhibitor | 345 | 341 | 686

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment
Description: Primary outcome was a composite of the development of referable diabetic retinopathy or referable maculopathy, or treatment for diabetic retinopathy or maculopathy (including retinal laser therapy, vitrectomy or intravitreal injection of medication). Referable diabetic retinopathy was defined by the NHS Scotland's grading criteria as any development of R3, R4 or M2 disease. R3 (referable background diabetic retinopathy): any of four or more blot hemorrhages in both inferior and superior hemi-fields, or venous beading, or intraretinal microvascular abnormalities (IRMA); R4 (proliferative diabetic retinopathy): any active new vessels, or vitreous hemorrhage; M2 (referable maculopathy): any blot hemorrhages, or hard exudates within a radius of ≤1 optic disc diameter of the centre of the fovea. Adverse event reports of eye procedures, vitreous haemorrhages and macular oedema were adjudicated by experienced doctors at the Central Co-ordinating Office (CCO), masked to treatment allocation.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: Intention-to-treat comparisons among all randomised participants of the effects of allocation to fenofibrate versus placebo during the scheduled treatment period on time to the first occurrence.
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 576 | 575
Participants | 131 | 168
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; Test type: Superiority — For the time-to-event analyses, survival analytic methods will be used to evaluate the time to the first event during the entire study period. Cox proportional hazards regression analyses, adjusted for baseline covariates used in minimised randomisation, will be used to estimate the hazard ratios, 95% confidence intervals and corresponding p-values, comparing all participants allocated active fenofibrate with all those allocated placebo; p = 0.006, Regression, Cox; Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.58 to 0.91]

2. Secondary Outcome: Number of Participants With the Individual Component of the Composite Primary Outcome: Development of Referable Diabetic Retinopathy or Maculopathy
Description: Progression of Diabetic Retinopathy/Maculopathy to a referable grade (R3 or R4 or M2) based on the NHS Scotland grading scheme in at least one eye.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 576 | 575
Participants | 130 | 168
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; Cox proportional hazards regression analyses were used to estimate the hazard ratio and 95% confidence intervals, comparing all participants allocated active fenofibrate with all those allocated placebo; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; p = 0.005, Regression, Cox; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.57 to 0.91]

3. Secondary Outcome: Number of Participants With the Individual Component of Composite Primary Outcome: Treatment for Diabetic Retinopathy or Maculopathy
Description: Treatment for diabetic retinopathy or maculopathy (including intravitreal injection of medication, retinal laser therapy, or vitrectomy) in either eye.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: Intention-to-treat comparisons among all randomised participants of the effects of allocation to fenofibrate versus placebo during the scheduled treatment period on time to first occurrence.
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 576 | 575
Participants | 17 | 28
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; p = 0.08, Regression, Cox; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.31 to 1.06]

4. Secondary Outcome: Number of Participants With Any Progression of Diabetic Retinopathy or Maculopathy Across the NHS Scotland Retinopathy Grading Scale
Description: Any progression of diabetic retinopathy or maculopathy across the NHS Scotland retinopathy grading scale. R4 = Proliferative DR, R3 = Referable background DR, R2 = Observable background DR. R1 = Mild background DR, R0 = No DR anywhere (where R4 is the highest severity grade and R0 is the lowest grade); M2 = Referable maculopathy, M1 = Observable maculopathy, M0 = No Maculopathy (where M2 is the highest severity grade and M0 is the lowest grade).
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 576 | 575
Participants | 185 | 231
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; p = 0.003, Regression, Cox; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.61 to 0.90]

5. Secondary Outcome: Number of Participants With Referable Maculopathy (Exudates or Blot Haemorrhages Within One Disc Diameter of the Fovea)
Description: The presence of hard exudates or blot haemorrhages within 1 disc diameter of the macula/fovea
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 576 | 575
Participants | 107 | 149
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; p = 0.001, Regression, Cox; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.52 to 0.85]

6. Secondary Outcome: Number of Participants With The Development of Macular Oedema
Description: The accumulation of macular fluid as determined by optical coherence tomography (OCT) imaging or on adverse event report
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 576 | 575
Participants | 22 | 43
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; p = 0.008, Regression, Cox; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.30 to 0.84]

7. Secondary Outcome: Visual Acuity
Description: Based on measurement of visual acuity at retinal screening visits. Baseline visual acuity was taken from routine measurement within NHS Scotland's Diabetic Eye Screening programme (using the latest value within 18 months of randomisation). Visual acuity after randomisation was obtained by averaging available results for a participant. Conversion from Snellen to LogMAR was applied where necessary. This analysis is based on the better eye: if only 1 eye with results, analyse that eye; if 2 eyes, use eye with better acuity; if identical acuity in both eyes, use the right eye. LogMAR typically ranges from -0.3 (20/10 vision on the Snellen chart) to 1 (20/200 vision). Lower scores indicate better vision.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: Intention-to-treat comparisons among all randomised participants of the effects of allocation to fenofibrate versus placebo during the scheduled treatment period on trial-averaged visual acuity.
Measure: Mean (95% Confidence Interval); unit: LogMAR
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 555 | 557
LogMAR | 0.06 [0.05 to 0.07] | 0.05 [0.05 to 0.06]
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; The estimates were derived from linear mixed model repeated measures; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation and for the baseline visual acuity; p = 0.36, Regression, Cox; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.01 to 0.01]

8. Secondary Outcome: Visual Function, Based on the National Eye Institute Visual Functioning Questionnaire 25 (VFQ-25).
Description: Visual function is based on the Visual Function Questionnaire-25. Visual function was defined by the composite score derived from the VFQ-25. VFQ-25 data were collected at the screening visit, after two years and at the end of the study. Results from two years and end-of-study were averaged to provide a trial-averaged result for a participant. The VFQ-25 composite score ranges from 0 to 100, where higher scores indicate better visual function. It is calculated by averaging results from up to 11 vision-related sub-scales.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: Intention-to-treat comparisons among all randomised participants of the effects of allocation to fenofibrate versus placebo during the scheduled treatment period on trial-averaged VFQ-25 Composite Score. Collected at baseline, at approximately 2 years and at the end of the trial.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 491 | 498
score on a scale | 90 [89 to 91] | 89 [89 to 90]
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; The estimates were derived from linear mixed model repeated measures; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation and for baseline VFQ-25 composite score; p = 0.58, Regression, Cox; Mean Difference (Final Values) = 0, 95% CI 2-sided [-1 to 1]

9. Secondary Outcome: Quality of Life, Based on the EQ-5D Index Score
Description: Quality of life was measured using the EQ-5D instrument, and valued by mapping to the EQ-5D-3L UK value set using the mapping function developed by Hernandez Alava et al. Pharmaco Economics (2022). EQ-5D data were collected at the screening visit, after two years and at the end of the study. Results from two years and end-of-study were averaged to provide a trial-averaged result for a participant. Possible scores range from -0.59 to 1.00, where 1 is the best possible health state and 0 represents a quality of life considered equivalent to death.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: Intention-to-treat comparisons among all randomised participants of the effects of allocation to fenofibrate versus placebo during the scheduled treatment period on trial-averaged EQ-5D Index Score. Collected at baseline, at approximately 2 years and at the end of the trial.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 490 | 495
score on a scale | 0.75 [0.73 to 0.76] | 0.75 [0.74 to 0.76]
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; The estimates were derived from linear mixed model repeated measures; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation and for baseline EQ-5D Index Score; p = 0.93, Regression, Cox; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.02 to 0.02]

10. Secondary Outcome: Quality of Life, Based on the EQ-5D Visual Analogue Scale.
Description: EQ-5D Visual Analogue Scale data were collected at the screening visit, after two years and at the end of the study. Results from two years and end-of-study were averaged to provide a trial-averaged result for a participant. EQ VAS scores range from 0 to 100, where 100 is the best possible health state.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: Intention-to-treat comparisons among all randomised participants of the effects of allocation to fenofibrate versus placebo during the scheduled treatment period on trial-averaged EQ-5D Visual Analogue Scale. Collected at baseline, at approximately 2 years and at the end of the trial.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 491 | 495
score on a scale | 75 [74 to 76] | 76 [75 to 77]
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; The estimates were derived from a linear mixed model repeated measures; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation and for baseline EQ-5D Visual Analogue Score; p = 0.43, Regression, Cox; Mean Difference (Final Values) = -1, 95% CI 2-sided [-2 to 1]

11. Secondary Outcome: Cost to the Health Service
Description: Health economic analysis: cost to the health service over 2 years. This included (i) hospital inpatient and outpatient activity (costed with nationally representative NHS costs); (ii) costs of fenofibrate (based on 200mg NHS cost); (iii) laboratory tests (NHS cost (including nurse/doctor time)); (iv) community prescribed medicines (NHS costs); (v) NHS Scotland retinal screening (published NHS unit costs); (vi) treatment for advanced retinopathy: for relevant participants, application of assumptions regarding usual number of injections from UK cohort study.
Time Frame: 2 years
Population: Comparisons among all randomised participants of the effects of allocation to fenofibrate versus placebo over 2 years
Measure: Mean (95% Confidence Interval); unit: GBP (British Pounds)
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 576 | 575
GBP (British Pounds) | 3566 [3088 to 4364] | 3820 [3052 to 4749]
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; Test type: Other; Mean Difference (Final Values) = -254, 95% CI 2-sided [-1062 to 624]

12. Secondary Outcome: Cost-effectiveness (Incremental Cost Per QALY Gained)
Description: Health economic analysis: Cost-effectiveness (incremental cost per QALY gained). The result is the value of GBP (British Pound) expenditure required to gain 1 quality adjusted life year for fenofibrate therapy vs. standard care. Years gained are presented by arm with 95% credible intervals taken as 2.5th and 97.5th percentile of simulated probabilistic output.
Time Frame: Projected over 10 year horizon
Population: QALY calculated based on quality of life data from EQ-5D questionnaires collected at baseline, at approximately 2 years and at the end of the trial.
Measure: Mean (95% Confidence Interval); unit: Years gained
Groups:
- Fenofibrate 145mg: Fenofibrate 145 mg: One tablet (taken daily with normal renal function, taken every second day with chronic kidney disease)
Arm/Group | Fenofibrate 145mg | Placebo Oral Tablet
Number analyzed (Participants) | 576 | 575
Years gained | 5.434 [5.332 to 5.540] | 5.419 [5.319 to 5.525]
Statistical Analysis 1: Comparison: Fenofibrate 145mg vs Placebo Oral Tablet; Test type: Other; Incremental cost-effectiveness ratio = 614 — £614 cost per QALY gained based on probabilistic analysis

13. Secondary Outcome: Number of Participants in Subgroup Sex - Male With Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment
Description: Composite primary outcome in prespecified subgroup according to the baseline characteristic: Sex - male. The primary outcome was a composite of the development of referable diabetic retinopathy, or treatment for diabetic retinopathy or maculopathy (including retinal laser therapy, vitrectomy or intravitreal injection of medication). The definition for referable diabetic retinopathy is provided above in '1. Primary Outcome: Number of Participants with Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 420 | 419
Participants | 99 | 121
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.58 to 0.99]

14. Secondary Outcome: Number of Participants in Subgroup Sex - Female With Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment
Description: Composite primary outcome in prespecified subgroup according to the baseline characteristic: Sex - female. The primary outcome was a composite of the development of referable diabetic retinopathy, or treatment for diabetic retinopathy or maculopathy (including retinal laser therapy, vitrectomy or intravitreal injection of medication). The definition for referable diabetic retinopathy is provided above in '1. Primary Outcome: Number of Participants with Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 156 | 156
Participants | 32 | 47
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.40 to 1.00]

15. Secondary Outcome: Number of Participants in Subgroup Age <60y With Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment
Description: Composite primary outcome in prespecified subgroup according to the baseline characteristic: Age <60 years. The primary outcome was a composite of the development of referable diabetic retinopathy, or treatment for diabetic retinopathy or maculopathy (including retinal laser therapy, vitrectomy or intravitreal injection of medication). The definition for referable diabetic retinopathy is provided above in '1. Primary Outcome: Number of Participants with Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 249 | 264
Participants | 68 | 93
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.52 to 0.97]

16. Secondary Outcome: Number of Participants in Subgroup Age ≥60y With Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment.
Description: Composite primary outcome in prespecified subgroup according to the baseline characteristic: Age ≥60 years. The primary outcome was a composite of the development of referable diabetic retinopathy, or treatment for diabetic retinopathy or maculopathy (including retinal laser therapy, vitrectomy or intravitreal injection of medication). The definition for referable diabetic retinopathy is provided above in '1. Primary Outcome: Number of Participants with Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 327 | 311
Participants | 63 | 75
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.55 to 1.07]

17. Secondary Outcome: Number of Participants in Subgroup - Type 1 Diabetes With Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment
Description: Composite primary outcome in prespecified subgroup according to the baseline characteristic: Type of Diabetes - type 1 diabetes. The primary outcome was a composite of the development of referable diabetic retinopathy, or treatment for diabetic retinopathy or maculopathy (including retinal laser therapy, vitrectomy or intravitreal injection of medication). The definition for referable diabetic retinopathy is provided above in '1. Primary Outcome: Number of Participants with Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 154 | 151
Participants | 38 | 45
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.51 to 1.21]

18. Secondary Outcome: Number of Participants in Subgroup - Type 2 or Other Type of Diabetes With Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment
Description: Composite primary outcome in prespecified subgroup according to the baseline characteristic: Type 2 and other diabetes. The primary outcome was a composite of the development of referable diabetic retinopathy, or treatment for diabetic retinopathy or maculopathy (including retinal laser therapy, vitrectomy or intravitreal injection of medication). The definition for referable diabetic retinopathy is provided above in '1. Primary Outcome: Number of Participants with Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 422 | 424
Participants | 93 | 123
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.54 to 0.93]

19. Secondary Outcome: Number of Participants in Subgroup - eGFR <60 mL/Min/1.73m^2 With Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment
Description: Primary outcome in prespecified subgroup according to the baseline characteristic: Renal function at Randomisation - eGFR <60mL/min/1.73m^2). The primary outcome was a composite of the development of referable diabetic retinopathy, or treatment for diabetic retinopathy or maculopathy (including retinal laser therapy, vitrectomy or intravitreal injection of medication). The definition for referable diabetic retinopathy is provided above in '1. Primary Outcome: Number of Participants with Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 130 | 131
Participants | 17 | 32
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.28 to 0.93]

20. Secondary Outcome: Number of Participants in Subgroup - eGFR ≥60 mL/Min/1.73m^2 With Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment
Description: Composite primary outcome in prespecified subgroup according to the baseline characteristic: Renal function at Randomisation - eGFR ≥60mL/min/1.73m^2. The primary outcome was a composite of the development of referable diabetic retinopathy, or treatment for diabetic retinopathy or maculopathy (including retinal laser therapy, vitrectomy or intravitreal injection of medication). The definition for referable diabetic retinopathy is provided above in '1. Primary Outcome: Number of Participants with Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 446 | 444
Participants | 114 | 136
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.60 to 0.99]

21. Secondary Outcome: Number of Participants in Subgroup - HbA1c <70 mmol/Mol With Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment
Description: Primary outcome in prespecified subgroup according to the baseline characteristic: HbA1c at Screening <70mmol/mol. The primary outcome was a composite of the development of referable diabetic retinopathy, or treatment for diabetic retinopathy or maculopathy (including retinal laser therapy, vitrectomy or intravitreal injection of medication). The definition for referable diabetic retinopathy is provided above in '1. Primary Outcome: Number of Participants with Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 361 | 346
Participants | 63 | 81
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.49 to 0.95]

22. Secondary Outcome: Number of Participants in Subgroup - HbA1c ≥70 mmol/Mol With Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment
Description: Primary outcome in prespecified subgroup according to the baseline characteristic-HbA1c at Screening - ≥70mmol/mol. The primary outcome was a composite of the development of referable diabetic retinopathy, or treatment for diabetic retinopathy or maculopathy (including retinal laser therapy, vitrectomy or intravitreal injection of medication). The definition for referable diabetic retinopathy is provided above in '1. Primary Outcome: Number of Participants with Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 177 | 193
Participants | 57 | 79
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.53 to 1.06]

23. Secondary Outcome: Number of Participants in Subgroup - HbA1c Unknown With Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment
Description: Composite primary outcome in prespecified subgroup according to the baseline characteristic - HbA1c at Screening - Unknown. The primary outcome was a composite of the development of referable diabetic retinopathy, or treatment for diabetic retinopathy or maculopathy (including retinal laser therapy, vitrectomy or intravitreal injection of medication). The definition for referable diabetic retinopathy is provided above in '1. Primary Outcome: Number of Participants with Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 38 | 36
Participants | 11 | 8
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 1.40, 95% CI 2-sided [0.55 to 3.57]

24. Secondary Outcome: Number of Participants in Subgroup With Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment, Within 1 Year of Randomization
Description: Composite primary outcome in prespecified subgroup according to the baseline characteristic: Timing of primary outcome - Within first year. The primary outcome was a composite of the development of referable diabetic retinopathy, or treatment for diabetic retinopathy or maculopathy (including retinal laser therapy, vitrectomy or intravitreal injection of medication). The definition for referable diabetic retinopathy is provided above in '1. Primary Outcome: Number of Participants with Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment.
Time Frame: Up to 1 year from randomisation.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 576 | 575
Participants | 45 | 63
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.48 to 1.03]

25. Secondary Outcome: Number of Participants in Subgroup With Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment, After 1 Year From Randomization
Description: Composite primary outcome in prespecified subgroup according to the baseline characteristic: Timing - After first year. The primary outcome was a composite of the development of referable diabetic retinopathy, or treatment for diabetic retinopathy or maculopathy (including retinal laser therapy, vitrectomy or intravitreal injection of medication). The definition for referable diabetic retinopathy is provided above in '1. Primary Outcome: Number of Participants with Progression to Referable Diabetic Retinopathy or Maculopathy, or Treatment.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years, excluding any primary outcome events within the first year of randomisation.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 525 | 509
Participants | 86 | 105
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.56 to 0.99]

26. Other Pre Specified Outcome: Percentage Change in Urine Albumin:Creatinine Ratio
Description: Based on collection of biochemical data. Urine albumin: creatinine ratio (UACR) results. Urine was collected for measurement of UACR at LENS screening visits wherever possible (baseline results). Post randomization UACR results came from measurements conducted part of routine care. Post randomisation results for a participant were averaged for each participant. Separate values for participants assigned fenofibrate and placebo are reported as geometric mean (95% confidence intervals) and the difference between arms is reported as a percentage difference (95% confidence intervals)
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: Intention-to-treat comparisons among randomised participants of the effects of allocation to fenofibrate versus placebo during the scheduled treatment period on trial-averaged UACR.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 462 | 474
mg/g | 13.6 [12.1 to 15.3] | 15.5 [13.8 to 17.5]
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; Linear mixed model repeated measures analyses were conducted to estimate the trial-averaged percentage difference in geometric mean UACR between the randomised treatment groups. UACR data at baseline was available for 312 participants allocated fenofibrate and 310 participants allocated placebo; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation and for the baseline UACR; Hazard Ratio (HR) = -12.4, 95% CI 2-sided [-25.8 to 3.5] — Estimates are in %

27. Other Pre Specified Outcome: Number of Participants With Occurrence of Major Cardiovascular Events (Myocardial Infarction, Stroke, Coronary or Peripheral Revascularisation)
Description: This outcome is a composite of myocardial infarction, stroke, coronary artery revascularisation and peripheral artery revascularisation.
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 576 | 575
Participants | 45 | 43
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.69 to 1.60]

28. Other Pre Specified Outcome: Number of Participants With Occurrence of Non-traumatic Lower Limb Amputations
Description: Composite of any non-traumatic lower limb amputation (defined as minor amputation [distal to the ankle] or major amputation [through or proximal to the ankle]).
Time Frame: 4.0 years (interquartile range, 3.6 to 4.3) years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
Number analyzed (Participants) | 576 | 575
Participants | 4 | 11
Statistical Analysis 1: Comparison: Fenofibrate 145 mg vs Placebo Oral Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Adjusted for baseline covariates used in minimised randomisation; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.11 to 1.12]

ADVERSE EVENTS:
Time Frame: 4 years
Description: Data collected were: (i) all deaths, (ii) all serious adverse events (AEs), (iii) all reasons for stopping study treatment (serious and non-serious AEs). It was pre-specified that it was only mandatory to record non-serious AEs if they led to cessation of study treatment. These are listed under 'Other AEs' below. AEs are reported according to MedDRA System Organ Class.
Arm/Group | Fenofibrate 145 mg | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 35/576 | 38/575
Serious Adverse Events (participants affected / at risk) | 208/576 | 204/575
Other Adverse Events (participants affected / at risk) | 17/576 | 21/575
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fenofibrate 145 mg (N=576) | Placebo Oral Tablet (N=575)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 5 | 2
Cardiac disorders (Cardiac disorders) | 37 | 36
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 0 | 0
Ear and labyrinth disorders (Ear and labyrinth disorders) | 0 | 0
Endocrine disorders (Endocrine disorders) | 1 | 1
Eye disorders (Eye disorders) | 6 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 21 | 27
General disorders and administration site conditions (General disorders) | 12 | 16
Hepatobiliary disorders (Hepatobiliary disorders) | 6 | 7
Immune system disorders (Immune system disorders) | 0 | 0
Infections and infestations (Infections and infestations) | 49 | 50
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 23 | 28
Investigations (Investigations) | 4 | 3
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 16 | 21
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 11 | 7
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 29 | 23
Nervous system disorders (Nervous system disorders) | 33 | 27
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 0 | 0
Psychiatric disorders (Psychiatric disorders) | 6 | 5
Renal and urinary disorders (Renal and urinary disorders) | 14 | 10
Reproductive system and breast disorders (Reproductive system and breast disorders) | 2 | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 19 | 14
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3 | 4
Social circumstances (Social circumstances) | 0 | 0
Surgical and medical procedures (Surgical and medical procedures) | 50 | 52
Vascular disorders (Vascular disorders) | 3 | 4
Product issues (Product Issues) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fenofibrate 145 mg (N=576) | Placebo Oral Tablet (N=575)
Eye disorders (Eye disorders) | 2 | 2 — It was not mandatory to record non-serious AEs unless they led to stopping study treatment. Only non-serious AEs leading to stopping study treatment are reported here.
Gastrointestinal disorders (Gastrointestinal disorders) | 6 | 5 — It was not mandatory to record non-serious AEs unless they led to stopping study treatment. Only non-serious AEs leading to stopping study treatment are reported here.
Hepatobiliary disorders (Hepatobiliary disorders) | 0 | 1 — It was not mandatory to record non-serious AEs unless they led to stopping study treatment. Only non-serious AEs leading to stopping study treatment are reported here.
Investigations (Investigations) | 1 | 3 — It was not mandatory to record non-serious AEs unless they led to stopping study treatment. Only non-serious AEs leading to stopping study treatment are reported here.
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 | 2 — It was not mandatory to record non-serious AEs unless they led to stopping study treatment. Only non-serious AEs leading to stopping study treatment are reported here.
Nervous system disorders (Nervous system disorders) | 4 | 3 — It was not mandatory to record non-serious AEs unless they led to stopping study treatment. Only non-serious AEs leading to stopping study treatment are reported here.
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — It was not mandatory to record non-serious AEs unless they led to stopping study treatment. Only non-serious AEs leading to stopping study treatment are reported here.
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — It was not mandatory to record non-serious AEs unless they led to stopping study treatment. Only non-serious AEs leading to stopping study treatment are reported here.
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 | 3 — It was not mandatory to record non-serious AEs unless they led to stopping study treatment. Only non-serious AEs leading to stopping study treatment are reported here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT03439345/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT03439345/SAP_001.pdf